CLINICAL TRIAL: NCT06995599
Title: Thoracic Duct Ligation and Postoperative Weight Loss in Obese Patients Undergoing Minimally Invasive Lung Surgery: A Pilot Exploratory Clinical Study
Brief Title: Impact of Thoracic Duct Ligation on Postoperative Weight Reduction in Obese Patients Receiving Minimally Invasive Lung Surgery: A Clinical Investigation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yongxin Zhou (Other)
Responsible Party: Sponsor-Investigator, Yongxin Zhou, Chief Surgeon, Department of Thoracic Surgery, Shanghai Tongji Hospital, Tongji University School of Medicine
Organization: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ethics Review No. 2025-003
Record Dates: First submitted 2025-04-02; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Obese Patients
Keywords: Obesity; therapy; Metabolic Effects of Thoracic Duct Ligation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Primary comparison: Preoperative (baseline) vs. postoperative parameters within the same cohort.
  Secondary comparison: Outcomes compared to historical controls (patients who underwent lung surgery without thoracic duct ligation).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thoracic Duct Ligation (TDL) (Experimental)
  Interventions: Procedure: Thoracic Duct Ligation (TDL)

INTERVENTIONS:
Procedure: Thoracic Duct Ligation (TDL) — Following the minimally invasive right-sided lung cancer resection, during mediastinal lymph node dissection, the posterior aspect of the azygos vein is identified. The mediastinal pleura is then longitudinally incised along the medial border of the azygos vein and posterior to the esophagus. Between the azygos vein and aorta, the thoracic duct is meticulously localized as a milky-white translucent structure measuring 2-3 mm in diameter. A 5-mm segment of the duct is carefully mobilized and double-clamped with vascular clips under direct thoracoscopic visualization. The surgical field is thoroughly inspected to confirm the absence of chylous leakage, and the procedure is concluded after standard closure and confirmation of hemostasis.

SUMMARY:
This clinical trial aims to investigate whether thoracic duct ligation (TDL) can improve obesity and lipid metabolism. The primary questions it seeks to answer are:

Whether thoracic duct ligation can improve BMI and lipid metabolism in obese patients.

The safety and feasibility of thoracic duct ligation as a treatment for obesity.

DETAILED DESCRIPTION:
Background:

Obesity (BMI≥28 kg/m²) is a global health crisis with limited effective interventions. Emerging evidence suggests that TDL-a routine step in esophagectomy-may reduce body weight and improve lipid profiles, but its therapeutic potential for metabolic modulation remains unexplored.

Objectives:

Primary: Assess safety and feasibility of TDL during video-assisted thoracoscopic surgery (VATS) for stage IA1-IB lung cancer with concurrent obesity (BMI≥30 kg/m²).

Secondary: Evaluate changes in body weight (%), lipid metabolism (LDL/HDL), inflammatory markers (CRP, IL-6), and fat-soluble vitamin levels.

Methods:

Single-center prospective cohort with longitudinal monitoring. Eligible patients will undergo VATS + TDL, with metabolic parameters measured preoperatively and at postoperative day 1/5, months 1/3/6/12.

Exploratory Endpoints:

* Weight loss trajectory (% total body weight)
* Mechanisms of metabolic reprogramming (e.g., gut hormone shifts)
* Procedure-related morbidity (lymphatic leakage, vitamin deficiency)

Significance:

First study to evaluate TDL as a potential metabolic therapy in non-esophageal surgery, providing preliminary data for future randomized trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age & Gender: Individuals aged 18-75 years, regardless of gender.
2. Clinical Profile:Diagnosed with early-stage lung cancer (stage IA1-IB) and obesity (BMI ≥28 kg/m²).
3. Scheduled to undergo video-assisted thoracoscopic surgery (VATS) for right-sided lung cancer resection at our institution between October 2024 and October 2026.
4. Surgical Eligibility: Approved for surgery following multidisciplinary team (MDT) assessment.
5. Treatment Plan: No requirement for adjuvant therapy post-lung resection.
6. Preoperative Evaluation:Completed standard preoperative workup, including:
7. Chest CT、Brain CT/MRI、Abdominal ultrasound OR PET-CT to rule out distant metastasis.
8. Informed Consent: Willing and able to comply with study requirements, with written informed consent provided.

Exclusion Criteria:

1. Concurrent Thoracic Infections: Patients with active intrathoracic infectious diseases (e.g., inflammatory conditions, tuberculosis).
2. Refusal of Novel Technique: Patients unwilling to undergo intraoperative thoracic duct ligation.
3. Clinically Unstable Comorbidities: Severe, unstable cardiovascular, renal, or respiratory disorders.
4. Prior Bariatric Surgery: History of weight-loss surgery (e.g., gastric bypass, sleeve gastrectomy).
5. Recent Trial Participation: Enrollment in other clinical trials within 30 days prior to screening.
6. Investigator Discretion: Other conditions deemed by the investigator to contraindicate participation.

Ages: 18 Days to 75 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Height and weight (for BMI calculation) | Height and weight (for BMI calculation) : Measured at baseline, postoperative 1/4/ 7/10/13/19/25/37months.;Lipid profile (LDL/HDL): Baseline, postoperative 1/5day, 1/4/ 7/10/13/19/25/37months.Participants will be followed for up to 36 months .
  Height and weight (for BMI calculation)

IPD SHARING:
Plan to Share IPD: No